CLINICAL TRIAL: NCT02569814
Title: A Study to Compare the Pharmacokinetics and Safety of a Fixed Dose Combination of Fimasartan/Amlodipine/Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FARC-CT-102
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — fimasartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Subjects of Group 1 take Fimasartan/Amlodipine Combination Tablet and Rosuvastatin Individual Tablets at 1st day as period I. And then, after wash out for 2 weeks, as period II, subjects of Group 1 take a Fimasartan/Amlodipine/Rosuvastatin Combination Tablet at 15th day.
  Interventions: Drug: Fimasartan/Amlodipine/Rosuvastatin; Drug: Fimasartan/Amlodipine; Drug: Rosuvastatin
- Group 2 (Other): Subjects of Group 2 take a Fimasartan/Amlodipine/Rosuvastatin Combination Tablet at 1st day as period I. And then, after wash out for 2 weeks, as period II, subjects of Group 2 take Fimasartan/Amlodipine Combination Tablet and Rosuvastatin Individual Tablets at 15th day.
  Interventions: Drug: Fimasartan/Amlodipine/Rosuvastatin; Drug: Fimasartan/Amlodipine; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Fimasartan/Amlodipine/Rosuvastatin
Drug: Fimasartan/Amlodipine
Drug: Rosuvastatin

SUMMARY:
A Open-label, Randomized, Single-dose, 2x2 Crossover Study to Compare the Pharmacokinetics and Safety between a Fixed Dose Combination of Fimasartan/Amlodipine/Rosuvastatin versus Co-administration of a Fixed Dose Combination of Fimasartan/Amlodipine and Rosuvastatin in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* a Healthy male subject, aged 19- 50 years

Exclusion Criteria:

* History of clinically significant hypersensitivity to study drug, any other drug
* Hypotension or hypertension
* Active liver disease
* History of gastrointestinal disease
* History of excessive alcohol abuse
* Participation in any other study within 3 months

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cmax of Fimasartan, Amlodipine and Rosuvastatin | 0~144 hour after medication
AUCt(Area Under the Curve) of Fimasartan, Amlodipine and Rosuvastatin | 0~144 hour after medication

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea